CLINICAL TRIAL: NCT00524810
Title: A Multi-center Phase II Study Evaluating the Efficacy and Tolerance of the Association of Liposomal Doxorubicin and Docetaxel in First Line Chemotherapy in Patients With Metastatic Breast Cancer
Brief Title: Liposomal Doxorubicin and Docetaxel in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Douglas Micheau, ARCAGY-GINECO
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPYTTOLE
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caelyx - Taxotere (Experimental)
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Docetaxel

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — Caelyx 30 mg/m² day 1 every 3 weeks
  Other Names: Caelyx
Drug: Docetaxel — Taxotere 75 mg/m² day 2 every 3 weeks
  Other Names: Taxotere

SUMMARY:
Evaluation of safety and efficacy of a treatment associating Pegylated Liposomal Doxorubicin + Docetaxel in patients with metastatic breast cancer

DETAILED DESCRIPTION:
Evaluation of safety and efficacy of a treatment associating Pegylated Liposomal Doxorubicin + Docetaxel in patients with metastatic breast cancer. Patients will receive pyridoxin to prevent cutaneo-mucinous toxicities.

ELIGIBILITY:
Inclusion Criteria:

* first metastatic chemo line
* presence of measurable or bone lesion
* at least one lesion outside the radiated areas
* can have previously received hormonotherapy, chemotherapy in adjuvant phase, radiotherapy if older than 4 weeks

Exclusion Criteria:

* only local tumoral progression
* symptomatic cerebral metastasis
* neuropathy > NCI-CTC 2
* previous cancer within 10 years _ previous cancer within 10 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Non-progression rate after 6 cycles | 6 months

SECONDARY OUTCOMES:
tolerance and toxicity | 6 months
Tumor response and duration | 5 years
Time to Progression | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laure CHAUVENET, MD, PHD, Principal Investigator — Hôpital HOTEL DIEU - Paris
Locations (1):
- Hôpital HOTEL DIEU, Paris, France